CLINICAL TRIAL: NCT02481141
Title: Prospective, Randomized, Single-Blind, Placebo-Controlled, Dose-Escalation Pilot Study to Evaluate the Safety and Efficacy of 5-ALA-SFC in Subjects With Type II Diabetes
Brief Title: Pilot Study to Evaluate the Safety and Efficacy of 5-ALA-SFC in Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SBI Pharmaceuticals Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBIP12-002F
Record Dates: First submitted 2015-06-17; First posted 2015-06-25 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-ALA-SFC (Active Comparator): Study product administration will be as follows:
  Beginning Week 0: 1 capsule of 50mg 5-ALA-SFC twice per day for 2 weeks Beginning Week 2: 1 capsule of 75mg 5-ALA-SFC twice per day for 2 weeks Beginning Week 4: 1 capsule of 100mg 5-ALA-SFC twice per day for 8 weeks
  Interventions: Drug: 5-ALA-SFC
- Placebo (Placebo Comparator): Study matching placebo administration will be as follows:
  Beginning Week 0: 1 capsule twice per day for 2 weeks Beginning Week 2: 1 capsule twice per day for 2 weeks Beginning Week 4: 1 capsule twice per day for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5-ALA-SFC — Study product will be in the form of white-opaque capsules for oral administration, containing either 50, 75, or 100 mg of active 5-ALA - SFC
  Arms: 5-ALA-SFC
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this pilot study is to assess the safety and preliminary efficacy of 5-ALA - SFC at doses up to 200 mg per day in subjects with type II diabetes.

DETAILED DESCRIPTION:
The primary objective is to assess the safety of 5-ALA - SFC at doses up to 200 mg per day in subjects with type II diabetes mellitus. Safety will be assessed by the incidence of adverse events and clinically significant laboratory results.

The secondary objective is to assess the efficacy of 5-ALA-SFC at doses up to 200 mg per day on glycemic control in subjects with type II diabetes mellitus. Efficacy measures will include fasting plasma glucose level, HbA1c level, lipid profile, and body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females residing in Bahrain aged 20 to 75 years old
2. Otherwise in good health in the opinion of the investigator based on results of medical history, physical exam and laboratory assessments
3. Diagnosed with type II diabetes mellitus with HbA1c >6.5 and <10% which is uncontrolled despite the use of one or more glycemia-lowering drugs
4. BMI ≤44 kg/m2
5. Sitting BP ≤ 160/100mm Hg
6. Sleep apnea screening is negative
7. Ophthalmological exam is within normal limits as judged by the investigator. If findings are observed, they must be judged as not clinically significant.
8. Female subjects are not pregnant, not breast-feeding, and if of childbearing potential, have agreed to use an acceptable method of birth control

Exclusion Criteria:

1. Liver dysfunction defined as liver function tests >1.5 times upper limit of normal
2. Renal dysfunction defined as BUN and/or serum creatinine >1.5 times upper limit of normal and/or eGFR <30 ml/min/1.73 m2
3. History of any life-threatening disease, cardiovascular disease, viral hepatitis, porphyria or hemochromatosis
4. Allergy to ALA, SFC, or any other component of study product
5. Use of insulin for management of serum glucose
6. Hypoglycemic event within the previous 3 months, defined as serum glucose levels less than 70 mg/dL
7. History of sickle cell anemia disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riyadh Rehani, Ph.D., Study Director — SBI Pharmaceuticals Co, Ltd.

REFERENCES:
- [Derived] Al-Saber F, Aldosari W, Alselaiti M, Khalfan H, Kaladari A, Khan G, Harb G, Rehani R, Kudo S, Koda A, Tanaka T, Nakajima M, Darwish A. The Safety and Tolerability of 5-Aminolevulinic Acid Phosphate with Sodium Ferrous Citrate in Patients with Type 2 Diabetes Mellitus in Bahrain. J Diabetes Res. 2016;2016:8294805. doi: 10.1155/2016/8294805. Epub 2016 Sep 22. PMID 27738640

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-ALA-SFC: Study product administration will be as follows:
  Beginning Week 0: 1 capsule of 50mg 5-ALA-SFC twice per day for 2 weeks Beginning Week 2: 1 capsule of 75mg 5-ALA-SFC twice per day for 2 weeks Beginning Week 4: 1 capsule of 100mg 5-ALA-SFC twice per day for 8 weeks
  5-ALA-SFC: Study product will be in the form of white-opaque capsules for oral administration, containing either 50, 75, or 100 mg of active 5-ALA - SFC
- Placebo: Study matching placebo administration will be as follows:
  Beginning Week 0: 1 capsule twice per day for 2 weeks Beginning Week 2: 1 capsule twice per day for 2 weeks Beginning Week 4: 1 capsule twice per day for 8 weeks
  Placebo
Period: Overall Study
Arm/Group | 5-ALA-SFC | Placebo
Started | 35 | 18
Completed | 26 | 13
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (ITT) included all patients who took at least one dose of study product and had at least one post-baseline efficacy evaluation
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-ALA-SFC | Placebo | Total
Number analyzed (Participants) | 35 | 15 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 15 | 48
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (6.51) | 51.9 (5.07) | 52.2 (6.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 33 | 13 | 46
Region of Enrollment [Number; unit: participants]
  Bahrain | 35 | 15 | 50

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Adverse Events as a Measure of Safety and Tolerability
Description: The objective of the current study was to investigate the safety and preliminary efficacy of doses up to 200 mg 5-ALA - SFC in a population of patients with type 2 diabetes mellitus living in Bahrain.
Time Frame: Week 2, Week 4, Week 12
Population: Safety population included all subjects who took at least one dose of study product.
Measure: Count of Participants; unit: Participants
Groups:
- 5-ALA-SFC Through Week 2 (50 mg 2x/Day): Study product administration will be as follows:
  Beginning Week 0: 1 capsule of 50mg 5-ALA-SFC twice per day for 2 weeks
- 5-ALA-SFC Through Week 4 (75 mg 2x/Day); 5-ALA-SFC Through Week 12 (100 mg 2x/Day): Study product administration will be as follows:
  Beginning Week 2: 1 capsule of 75mg 5-ALA-SFC twice per day for 2 weeks
- Placebo Through Week 2: Study matching placebo administration will be as follows:
  Beginning Week 0: 1 capsule twice per day for 2 weeks
- Placebo Through Week 4: Study matching placebo administration will be as follows:
  Beginning Week 2: 1 capsule twice per day for 2 weeks
- Placebo Through Week 12: Study matching placebo administration will be as follows:
  Beginning Week 4: 1 capsule twice per day for 8 weeks
Arm/Group | 5-ALA-SFC Through Week 2 (50 mg 2x/Day) | 5-ALA-SFC Through Week 4 (75 mg 2x/Day) | 5-ALA-SFC Through Week 12 (100 mg 2x/Day) | Placebo Through Week 2 | Placebo Through Week 4 | Placebo Through Week 12
Number analyzed (Participants) | 35 | 35 | 35 | 18 | 18 | 18
Participants | 6 | 8 | 2 | 3 | 1 | 1

2. Primary Outcome: Change From Baseline in Fasting Blood Glucose
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4, Week 12
Population: Intent-to-Treat Population (ITT) included all subjects who took at least one dose of study product and had at least one post-baseline efficacy evaluation. Change from Baseline was calculated as the mean for the visit compared to baseline mean for only the subjects with a result for that visit.
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- 5-ALA-SFC Through Week 2 (50 mg 2x/Day) Change From Baseline: Study product administration will be as follows:
  Beginning Week 0: 1 capsule of 50mg 5-ALA-SFC twice per day for 2 weeks
- 5-ALA-SFC Through Week 4 (75 mg 2x/Day) Change From Baseline: Study product administration will be as follows:
  Beginning Week 2: 1 capsule of 75mg 5-ALA-SFC twice per day for 2 weeks
- 5-ALA-SFC Through Wk 12 (100 mg 2x/Day) Change From Baseline: Study product administration will be as follows:
  Beginning Week 4: 1 capsule of 100mg 5-ALA-SFC twice per day for 8 weeks
- Placebo Through Week 2 Change From Baseline: Study matching placebo administration will be as follows:
  Beginning Week 0: 1 capsule twice per day for 2 weeks
- Placebo Through Week 4 Change From Baseline: Study matching placebo administration will be as follows:
  Beginning Week 2: 1 capsule twice per day for 2 weeks
- Placebo Through Week 12 Change From Baseline: Study matching placebo administration will be as follows:
  Beginning Week 4: 1 capsule twice per day for 8 weeks
Arm/Group | 5-ALA-SFC Through Week 2 (50 mg 2x/Day) Change From Baseline | 5-ALA-SFC Through Week 4 (75 mg 2x/Day) Change From Baseline | 5-ALA-SFC Through Wk 12 (100 mg 2x/Day) Change From Baseline | Placebo Through Week 2 Change From Baseline | Placebo Through Week 4 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 33 | 30 | 22 | 14 | 14 | 12
mg/dL | 2.3 (3.4) | -0.2 (4.9) | -3.0 (4.4) | -7.3 (5.2) | -0.8 (7.2) | -4.2 (5.9)

3. Secondary Outcome: Change From Baseline in 2 Hour Post Meal Glucose Level
Description: Change from baseline in blood glucose levels 2 hours after breakfast
Time Frame: Baseline, Week 2, Week 4, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- 5-ALA-SFC Through Week 12 (100 mg 2x/Day) Change From Baseline: Study product administration will be as follows:
  Beginning Week 4: 1 capsule of 100mg 5-ALA-SFC twice per day for 8 weeks
Arm/Group | 5-ALA-SFC Through Week 2 (50 mg 2x/Day) Change From Baseline | 5-ALA-SFC Through Week 4 (75 mg 2x/Day) Change From Baseline | 5-ALA-SFC Through Week 12 (100 mg 2x/Day) Change From Baseline | Placebo Through Week 2 Change From Baseline | Placebo Through Week 4 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 33 | 30 | 21 | 14 | 12 | 10
mg/dL | -0.2 (5.1) | -12.9 (6.1) | -8.5 (9.8) | -26.5 (7.8) | -18.8 (9.9) | -33.0 (14.2)

4. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline measured at week 6 and week 12 only
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: kg
Groups:
- 5-ALA-SFC Through Week 6 Change From Baseline: Week 6: 1 capsule of 100mg 5-ALA-SFC twice per day
- 5-ALA-SFC Through Week 12 Change From Baseline: Week 12: 1 capsule of 100mg 5-ALA-SFC twice per day
- Placebo Through Week 6 Change From Baseline: Week 6: 1 placebo capsule twice per day
- Placebo Through Week 12 Change From Baseline: Week 12: 1 placebo capsule twice per day
Arm/Group | 5-ALA-SFC Through Week 6 Change From Baseline | 5-ALA-SFC Through Week 12 Change From Baseline | Placebo Through Week 6 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 30 | 26 | 13 | 13
kg | -0.1 (0.5) | -0.2 (0.3) | -0.3 (0.7) | -0.8 (0.4)

5. Secondary Outcome: Change From Baseline in HbA1c
Description: Change from baseline in HbA1c %
Time Frame: Baseline, Week 2, Week 4, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of HbA1c
Groups:
- 5-ALA-SFC Through 4 (75 mg 2x/Day) Change From Baseline: Study product administration will be as follows:
  Beginning Week 2: 1 capsule of 75mg 5-ALA-SFC twice per day for 2 weeks
- 5-ALA-SFC Through 12 (100 mg 2x/Day) Change From Baseline: Study product administration will be as follows:
  Beginning Week 4: 1 capsule of 100mg 5-ALA-SFC twice per day for 8 weeks
Arm/Group | 5-ALA-SFC Through Week 2 (50 mg 2x/Day) Change From Baseline | 5-ALA-SFC Through 4 (75 mg 2x/Day) Change From Baseline | 5-ALA-SFC Through 12 (100 mg 2x/Day) Change From Baseline | Placebo Through Week 2 Change From Baseline | Placebo Through Week 4 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 32 | 30 | 25 | 13 | 13 | 13
percentage of HbA1c | -0.2 (0.1) | -0.3 (0.1) | -0.7 (0.2) | -0.5 (0.2) | -0.5 (0.2) | -0.5 (0.2)

6. Secondary Outcome: Change From Baseline in Total Cholesterol (Component of Lipid Profile)
Description: Change from baseline measured at week 6 and week 12 only
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5-ALA-SFC Through Week 6 Change From Baseline | 5-ALA-SFC Through Week 12 Change From Baseline | Placebo Through Week 6 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 27 | 25 | 13 | 13
mg/dL | -5.2 (3.7) | 6.8 (3.5) | -7.6 (5.5) | -0.1 (5.0)

7. Secondary Outcome: Change From Baseline LDL (Component of Lipid Profile)
Description: Change from baseline measured at week 6 and week 12 only
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5-ALA-SFC Through Week 6 Change From Baseline | 5-ALA-SFC Through Week 12 Change From Baseline | Placebo Through Week 6 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 27 | 25 | 13 | 13
mg/dL | -2.9 (3.2) | 7.6 (3.3) | -11.8 (4.7) | -4.0 (4.6)

8. Secondary Outcome: Change From Baseline in HDL (Component of Lipid Profile)
Description: Change from baseline measured at week 6 and week 12 only
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5-ALA-SFC Through Week 6 Change From Baseline | 5-ALA-SFC Through Week 12 Change From Baseline | Placebo Through Week 6 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 27 | 25 | 13 | 13
mg/dL | -0.8 (1.0) | 0.5 (1.0) | -1.6 (1.4) | -1.1 (1.4)

9. Secondary Outcome: Change From Baseline in Triglycerides (Component of Lipid Profile)
Description: Change from baseline measured at week 6 and week 12 only
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 5-ALA-SFC Through Week 6 Change From Baseline | 5-ALA-SFC Through Week 12 Change From Baseline | Placebo Through Week 6 Change From Baseline | Placebo Through Week 12 Change From Baseline
Number analyzed (Participants) | 27 | 25 | 13 | 13
mg/dL | -1.3 (14.6) | 3.2 (11.1) | 4.5 (21.1) | 11.9 (15.4)

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected during the 12 week period subjects were in the study and taking either 5-ALA-SFC or Placebo.
Groups:
- 5-ALA-SFC Through Week 2: Beginning Week 0: 1 capsule of 50mg 5-ALA-SFC twice per day for 2 weeks
- 5-ALA-SFC Through Week 4: Beginning Week 2: 1 capsule of 75mg 5-ALA-SFC twice per day for 2 weeks
- 5-ALA-SFC Through Week 12: Beginning Week 4: 1 capsule of 100mg 5-ALA-SFC twice per day for 8 weeks
- Placebo Through Week 2: Beginning Week 0: 1 placebo capsule twice per day for 2 weeks
- Placebo Through Week 4: Beginning Week 2: 1 placebo capsule twice per day for 2 weeks
- Placebo Through Week 12: Beginning Week 4: 1 placebo capsule twice per day for 8 weeks
Arm/Group | 5-ALA-SFC Through Week 2 | 5-ALA-SFC Through Week 4 | 5-ALA-SFC Through Week 12 | Placebo Through Week 2 | Placebo Through Week 4 | Placebo Through Week 12
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/35 | 0/35 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 6/35 | 14/35 | 16/35 | 3/18 | 4/18 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-ALA-SFC Through Week 2 (N=35) | 5-ALA-SFC Through Week 4 (N=35) | 5-ALA-SFC Through Week 12 (N=35) | Placebo Through Week 2 (N=18) | Placebo Through Week 4 (N=18) | Placebo Through Week 12 (N=18)
Abscess in the nose (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One serious adverse event of a nasal abscess requiring hospitalization was reported by a subject receiving 5-ALA-SFC, which was not related to study product.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-ALA-SFC Through Week 2 (N=35) | 5-ALA-SFC Through Week 4 (N=35) | 5-ALA-SFC Through Week 12 (N=35) | Placebo Through Week 2 (N=18) | Placebo Through Week 4 (N=18) | Placebo Through Week 12 (N=18)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No